CLINICAL TRIAL: NCT02154633
Title: Development of a Family Communication and Decision-support Intervention for Women That Carry a BRCA1 or a BRCA2 Mutation and Their At-Risk Female Family Members
Brief Title: Lessons Learned From the Family Gene Toolkit
Acronym: FGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RWJ68039; Nurse Faculty Scholar 68039 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Women With BRCA 1 or BRCA 2 Mutation; Non-tested Female Family Members

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Gene Toolkit (Experimental): Psychosocial educational presentations over the Internet (Webinars) Two Webinars lasting 1 hour each One follow-up phone call lasting 20 minutes
  Interventions: Behavioral: Family Gene Toolkit
- Delayed Family Gene Toolkit (Active Comparator): Psychosocial educational presentations over the Internet (Webinars) Two Webinars lasting 1 hour each One follow-up phone call lasting 20 minutes
  Interventions: Behavioral: Delayed Family Gene Toolkit

INTERVENTIONS:
Behavioral: Family Gene Toolkit — Psychosocial educational presentations over the Internet (Webinars) Two Webinars lasting 1 hour each One follow-up phone call lasting 20 minutes Webinars and phone calls are delivered to one mutation carrier and one non-tested relative Genetic counselors and nurses with master's degree and experienced in oncology deliver the content of the intervention
  Arms: Family Gene Toolkit
Behavioral: Delayed Family Gene Toolkit — Psychosocial educational presentations over the Internet (Webinars) Two Webinars lasting 1 hour each One follow-up phone call lasting 20 minutes Webinars and phone calls are delivered to one mutation carrier and one non-tested relative Genetic counselors and nurses with master's degree and experienced in oncology deliver the content of the intervention
  Arms: Delayed Family Gene Toolkit

SUMMARY:
Mutations in the BRCA1/2 genes are the primary cause of hereditary breast/ovarian cancer syndrome. Genetic testing identifies mutation carriers and enables them to manage their cancer risk (i.e. chemoprevention, risk-reducing surgery, or intensive surveillance). However, uptake of genetic testing among at-risk individuals is low, implying that information about the disease and genetic testing is not being communicated effectively among family members. Mutation carriers are distressed about disclosing test results, while their relatives do not understand the implications of a positive test result for their own health. Thus, interventions that support family communication about genetic risk, and address psychological distress of family members could contribute to more effective management of hereditary breast/ovarian cancer.

The project aims to develop a family communication and decision-support intervention to 1) increase family communication about BRCA1/2 mutations; 2) reduce psychological distress associated with these mutations; and 3) increase informed decision-making regarding uptake of BRCA1/2 testing among at-risk family members. Focus groups with mutation carriers and at-risk relatives will inform the refinement of the intervention, as well as timing and mode of delivery. Two group, pre-post test study with a new sample of mutation carriers and family members will be used to test the feasibility, acceptability, and effect of the intervention.

ELIGIBILITY:
Inclusion Criteria for mutation carrier:

1. had genetic testing for BRCA 1 or BRCA 2, and received positive test results;
2. are older than 18 years;
3. speak English;
4. agree to invite in the study one female relative who has ≥10% of carrying a genetic mutation AND did not have genetic testing; and
5. have access to an Internet enabled computer.

Inclusion Criteria for relatives

1. did not have genetic testing for BRCA 1 or BRCA 2;
2. are older than 18 years;
3. speak English; and
4. have access to an Internet enabled computer.

Exclusion Criteria:

* Women who have no female relatives
* Women who are unable to consent
* Women who do not have access to the Internet or the computer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2014-08-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Intention for genetic testing | 1 month post-intervention
  Intention to have genetic testing
Decisional conflict for genetic testing | 1 month post-intervention
  Difficulty deciding about having genetic testing
Decisional regret | 1 month post-intervention
  Regret after having genetic testing

SECONDARY OUTCOMES:
Knowledge of BRCA1/2 genetics | 1 month post-intervention
  Genetic literacy

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Katapodi, PhD, Principal Investigator — Adjunct Associate Professor w/ Tenure
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Request for data, explanation of research question, and time frame

REFERENCES:
- [Result] Katapodi MC, Jung M, Schafenacker AM, Milliron KJ, Mendelsohn-Victor KE, Merajver SD, Northouse LL. Development of a Web-based Family Intervention for BRCA Carriers and Their Biological Relatives: Acceptability, Feasibility, and Usability Study. JMIR Cancer. 2018 Apr 13;4(1):e7. doi: 10.2196/cancer.9210. PMID 29653920